CLINICAL TRIAL: NCT03353883
Title: Is Early Preparation With GnRh Agonists Injection on D-1 of Menses of Hormonal Replacement Cycle Improves Pregnancy Rate in Women With Impaired Ovulation and Undergoing Frozen-Thawed Embryo Transfer? A Randomized Controlled Study
Brief Title: Early Preparation With Gonadotropin- Releasing Hormon (GnRh) Agonists Injection With Frozen-Thawed Embryo Transfer?
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid mohammed salama, assistent professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: khalid 5
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group A) Midluteal Triptorelin depot (Active Comparator): infertile women with impaired ovulation who will be subjected to Triptorelin sustained release(Decapeptyl depot 375 mg one injection )at D-21 of previous menstrual cycle Hormon Replacement Therapy (HRT)Cyclo-Progynova (estradiol, norgestrel)(Group A). All patients received the same luteal support in the form of intravaginal progesterone two day before embryos transfer until blood pregnancy test was performed 14 days later. The classic Testart slow freezing and rapid thawing protocol was applied on stage-2 PN embryos. Endometrial thickness was measured in the midsagittal plane using transvaginal ultrasound (TVU). Clinical pregnancy was diagnosed by measurement of β-HCG level and was confirmed 2-weeks later by TVU.
  Interventions: Drug: Triptorelin SR
- (Group B)first day Triptorelin depot (Active Comparator): infertile women with impaired ovulation who will be subjected toTriptorelin sustained release(Decapeptyl depot 375 mg one injection) at D-1 of menses then Cyclo-Progynova (estradiol, norgestrel) (Group B). All patients received the same luteal support in the form of intravaginal progesterone two day before embryos transfer until blood pregnancy test was performed 14 days later. The classic Testart slow freezing and rapid thawing protocol was applied on stage-2 PN embryos. Endometrial thickness was measured in the midsagittal plane using transvaginal ultrasound (TVU). Clinical pregnancy was diagnosed by measurement of β-Human Chorionic Gonadotropin level and was confirmed 2-weeks later by TVU.
  Interventions: Drug: Triptorelin SR

INTERVENTIONS:
Drug: Triptorelin SR — GnRH agonist depot( Decapeptyl) will be taken in the previous mid luteal cycle in group A and the first day in group B
  Other Names: Decapeptyl

SUMMARY:
The study intended to include >200 infertile women with impaired ovulation who will be subjected to HRT at D-21 of previous menstrual cycle (Group A) or D-1 of menses of replacement cycle (Group B). All patients received the same luteal support in the form of intravaginal progesterone two day before embryos transfer until blood pregnancy test was performed 14 days later. Clinical pregnancy was diagnosed by measurement of β-human chorionic gonadotropin level and was confirmed 2-weeks later by TVU.

DETAILED DESCRIPTION:
The study intended to include >200 infertile women with impaired ovulation who will be subjected to HRT at D-21 of previous menstrual cycle (Group A) or D-1 of menses of replacement cycle (Group B). All patients received the same luteal support in the form of intravaginal progesterone two day before embryos transfer until blood pregnancy test was performed 14 days later. The classic Testart slow freezing and rapid thawing protocol was applied on stage-2 pronuclear embryos. Endometrial thickness was measured in the midsagittal plane using transvaginal ultrasound (TVU). Clinical pregnancy was diagnosed by measurement of β-human chorionic gonadotropin level and was confirmed 2-weeks later by TVU.

ELIGIBILITY:
Inclusion Criteria:infertile women with impaired ovulation -

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
pregnancy outcome | 4 weeks
  pregnancy test-Transvaginal sonograghy

CONTACTS AND LOCATIONS:
Overall Officials: Khalid M Salama, MD, Principal Investigator — Associate professor of obestetric and gynecology
Locations (1):
- Benha university hospital, Banhā, Qaluibia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Azimi Nekoo E, Chamani M, Shahrokh Tehrani E, Hossein Rashidi B, Davari Tanha F, Kalantari V. Artificial Endometrial Preparation for Frozen-Thawed Embryo Transfer with or without Pretreatment with Depot Gonadotropin Releasing Hormone Agonist in Women with Regular Menses. J Family Reprod Health. 2015 Mar;9(1):1-4. PMID 25904960
- See also: infertility — http://bu.edu.eg